CLINICAL TRIAL: NCT01311765
Title: Comparison of Two Durations of Antibiotic Therapy in the Treatment of Severe Postoperative Peritonitis Admitted in Intensive Care Unit: a Randomised Multicentre Study
Brief Title: Duration of Antibiotic Therapy in the Treatment of Severe Postoperative Peritonitis Admitted in ICU
Acronym: DURAPOP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P081248
Record Dates: First submitted 2011-02-22; First posted 2011-03-10 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-07

CONDITIONS: Postoperative Peritonitis
Keywords: Postoperative peritonitis; Intra-abdominal infection; Surgery; Laparotomy; Nosocomial infection; Antibiotic therapy; Duration of treatment; Multidrug resistant bacteria
MeSH Terms: conditions — Intraabdominal Infections; Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 8 day-antibiotherapy (Active Comparator): Duration of antibiotic therapy limited to 8 days: Antibiotics received for up to 8 days following surgery for postoperative peritonitis in patients hospitalised in intensive care unit
  Interventions: Other: Duration of antibiotic therapy limited to 8 days
- 15 day-antibiotherapy (No Intervention): Antibiotics received for up to15 days following surgery for postoperative peritonitis in patients hospitalised in intensive care unit corresponding to usual practice and recommendations

INTERVENTIONS:
Other: Duration of antibiotic therapy limited to 8 days — Initiation of adequate empiric antibiotics for postoperative peritonitis within 24 hours after surgery and up to 8 days. At randomisation performed on day 8, the patients assigned to the 8-day group (short-course group) stop their treatment
  Arms: 8 day-antibiotherapy

SUMMARY:
The investigators purpose is to demonstrate that a short antibiotic therapy (8 days) for postoperative peritonitis brings an increased number of antibiotic-free days over a 28 days period when compared to conventional (15 days) treatment.

DETAILED DESCRIPTION:
This is a prospective randomized study involving 25 centers. Our goal is to demonstrate in the course of postoperative peritonitis that a short antibiotic therapy (8 days) compared to conventional antibiotic treatment (15 days) decreases the duration of exposure to antibiotics over a 28 days period . Patients admitted in ICU, operated for postoperative peritonitis and receiving an adequate antibiotic therapy will be identified and after informed consent is obtained will be randomized to receive a short course of antibiotic therapy (8 days) or a long course of antibiotic therapy (15 days). The primary endpoint is the number of antibiotic-free days at D28 after inclusion (analysis of superiority) . Secondary endpoints include mortality at D45 after inclusion (analysis of equivalence), the occurrence of relapse of infection, success rate of clinically and microbiologically evaluable patients, and emergence of multidrug resistant microorganisms in clinical isolates or hygiene samples. Patient data through day 45 following the initial intervention or until hospital discharge will be tracked.

ELIGIBILITY:
Inclusion Criteria:

The eligible patients have to fulfill all the following criteria

1. patients admitted in intensive care unit
2. in the 24 hours following surgery for postoperative intra-abdominal infection (defined as gross pus or purulent effusion within the peritoneal cavity or in one or several collections). Postoperative infection will be defined as an infection observed in a delay of 60 days following a procedure (endoscopy, surgery (abdominal, urologic, gynecologic or vascular surgery or any surgery performed in the peritoneal or retroperitoneal space) or interventional radiology)
3. having peroperative microbiologic samples collected
4. receiving an empiric antibiotic therapy initiated within the first 24 hours after completion of surgery
5. with a written informed consent from the patient or the relative or the legal representative or with an emergency consent

Non-inclusion criteria :

Patients with one of the following criteria are eligible for the study :

1. age<18
2. pregnancy
3. Duration of stay following inclusion <72 hours
4. neutropenia (PMN<500/mm3) due to chemotherapy or hematological disease
5. AIDS stage C
6. Immunosuppressive therapy or prolonged steroid therapy (≥0.5 mg/kg/d of prednisone or equivalent >1 month
7. Bowel perforation following endoscopy treated in a delay <6 hours after injury
8. Uterine perforation following a surgical procedure treated in a delay <6 hours after injury
9. Moribund patient (SAPS II score >65 within 12 hours preceding inclusion)
10. Limitation of treatment previously decided
11. Surgery considered as non curative by the surgeon
12. Patient included in another clinical trial evaluating an antimicrobial agent

Secondary exclusion criteria:

Among the eligible patients, those who have one of the following criteria will be excluded

1. Negative culture of the peritoneal fluid
2. Peritoneal culture exclusively fungal
3. Inadequate empiric antibiotic therapy (not targeting all the microorganisms cultured from peritoneal or blood cultures) within 24 hours after surgery
4. Death between D1 and D8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2011-05; Primary Completion 2015-03 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The number of antibiotic-free days at D28 after inclusion | 28 days
  The number of antibiotic-free days at D28 after inclusion (analysis of superiority)

SECONDARY OUTCOMES:
Mortality at D45 after inclusion | 45 days
  Mortality at D45 after inclusion (analysis of equivalence)
Duration of ICU and hospital stay | 45 days
  Duration of ICU and hospital stay
Changes in SOFA score | 8 days
  Changes in SOFA score
Number of days alive without organ failure | 28 days
  Number of days alive without organ failure
Failure rate for clinically evaluable patients | 28 days
  Failure rate for clinically evaluable patients
Failure rate for microbiologically evaluable patients | 28 days
  Failure rate for microbiologically evaluable patients
Rate of relapse within 45 days | 45 days
  Rate of relapse within 45 days
Emergence of multidrug resistant microorganisms in clinical isolates and hygiene samples | ICU discharge
  Emergence of multidrug resistant microorganisms in clinical isolates and hygiene samples
Total cost of antibiotic agents | 28 days
  Total cost of antibiotic agents
Evolution of procalcitonin plasma concentration | 15 days
  Evolution of procalcitonin plasma concentration
Rate of death within 45 days in specific subpopulations (elderly patients >80 years ; morbidly obese patients BMI>25kg/m2 ; severe infection with SAPSII score >40 ;peritoneal infection involving pseudomonas or enterococci ; bacteriemic infections) | 45 days
  Rate of death within 45 days in specific subpopulations (elderly patients >80 years ; morbidly obese patients BMI>25kg/m2 ; severe infection with SAPSII score >40 ;peritoneal infection involving pseudomonas or enterococci ; bacteriemic infections)
Total cost of hospital stay and evaluation of costs and resources impact for the hospital administration | Hospital discharge
  Total cost of hospital stay and evaluation of costs and resources impact for the hospital administration

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Montravers, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bichat, Paris, France

REFERENCES:
- [Derived] Montravers P, Tubach F, Lescot T, Veber B, Esposito-Farese M, Seguin P, Paugam C, Lepape A, Meistelman C, Cousson J, Tesniere A, Plantefeve G, Blasco G, Asehnoune K, Jaber S, Lasocki S, Dupont H; DURAPOP Trial Group. Short-course antibiotic therapy for critically ill patients treated for postoperative intra-abdominal infection: the DURAPOP randomised clinical trial. Intensive Care Med. 2018 Mar;44(3):300-310. doi: 10.1007/s00134-018-5088-x. Epub 2018 Feb 26. PMID 29484469